CLINICAL TRIAL: NCT04464083
Title: Intraocular Pressure Measurements Using Ocular Response Analyzer After Accelerated Corneal Collagen Crosslinking With Riboflavin and Ultraviolet A in Keratoconus
Brief Title: IOP Measurements Using ORA After ACXL in Keratoconus
Status: Completed | Type: Observational
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Omar Said, Assistant professor of ophthalmology, Fayoum University
Other Study IDs: R110
Record Dates: First submitted 2020-07-05; First posted 2020-07-09 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: IOP Readings Before and After Accelerated Corneal Collagen Crosslinking (CXL)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: IOP Measurment — To determine IOP readings before and after accelerated corneal collagen crosslinking (CXL)

SUMMARY:
The investigators measured IOP by Goldmann applanation tonometry(GAT) before and 6 months after accelerated 8 minutes CXL in using Avedro Kxl ,and correlated with corneal resistance factor(CRF)using ORA, AC angle and CCT using Scheimpflug imaging.

ELIGIBILITY:
Inclusion Criteria:

* KC patient indicated for CXL

Exclusion Criteria:

* Advanced KC Glaucoma patients

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: all patients with KC and indicated for CXL
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-04-12 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
To determine IOP readings before and after accelerated corneal collagen crosslinking | April-October 2020

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum University, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
approval from the principal investigator